CLINICAL TRIAL: NCT04903769
Title: Stress Management and Resiliency Training Program for Parkinson's Disease Patients and Their Caregivers (SMART-PD)
Brief Title: Stress Management and Resiliency Training Program for Parkinson's Disease
Acronym: SMART-PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Parkinson's Disease Foundation (Other)
Responsible Party: Principal Investigator, Adam Gonzalez, Associate Professor of Psychiatry & Behavioral Health, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 663519
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: All participants will receive the SMART-PD intervention and will take baseline and follow-up assessments to determine the impact of the program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's Patients and Caregivers (Other): Will participate in the 8-session SMART-PD program as a participant with Parkinson's disease or as a caregiver of a participant with Parkinson's disease
  Interventions: Behavioral: Stress Management and Resiliency Training Program for Parkinson's Disease (SMART-PD)

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training Program for Parkinson's Disease (SMART-PD) — SMART-PD is a manualized intervention that teaches cognitive-behavioral techniques and relaxation skills to help participants learn to elicit the relaxation response, alter cognitive appraisals, improve healthy lifestyle behaviors (i.e., sleep, nutrition, physical activity) and access social support.

SUMMARY:
SMART-PD is an 8-session program designed to decrease the physiological, emotional, cognitive and behavioral effects of stress in participants with Parkinson's disease and their caregivers by teaching cognitive-behavioral techniques and relaxation skills to help participants learn to elicit the relaxation response, alter cognitive appraisals, improve healthy lifestyle behaviors and access social support. The SMART program has been shown to be effective for reducing mental health symptoms such as depression and anxiety as well as physical symptoms such as pain and in promoting positive health behaviors.

DETAILED DESCRIPTION:
This is an interventional study sponsored by the Parkinson's Foundation designed to measure the feasibility, acceptability, and initial impact of the SMART-PD program on participants with a recent (less than five years) diagnosis of Parkinson's disease and their caregivers. This program provides information and tools to help patients and their caregivers cope with the new PD diagnosis and manage the stress and negative mental health symptoms (such as anxiety and depression) associated with the diagnosis.

SMART-PD is a manualized 8-week intervention that teaches cognitive-behavioral techniques and relaxation skills to help participants learn to elicit the relaxation response, alter cognitive appraisals, improve healthy lifestyle behaviors (i.e., sleep, nutrition, physical activity) and access social support.

Participants will take baseline and follow-up questionnaires to ascertain the impact of the program on outcomes such as quality of life, emotional health, coping skills, and healthy lifestyle behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease within the past three years or caregiver of someone with a recent diagnosis of Parkinson's disease
* Ability to participate in 8 weekly program sessions via Microsoft Teams or in-person (as available)
* Ability to provide informed consent

Exclusion Criteria:

* Previous participation in the SMART program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment and participation | One year
  The number of participants who enroll and fully participate in the program will be used to measure the feasibility of using SMART-PD for patients with Parkinson's disease and their caregivers.
SMART Group Feedback Form | Eight weeks
  Designed to assess the accessibility of the SMART-PD program, The SMART Group Feedback form contains six Likert-scale questions such as, "On a 10-point scale, how would you rate the following items: helpfulness/effectiveness of SMART group" and four open-ended questions such as, "What has been the most helpful part of the group for you?"
Change from Baseline General Quality of Life at 1-week post-intervention | 1-week post-intervention
  The Short Form Health Survey (SF-36) is a quality of life measure that assesses eight aspects of health through the use of 36 multiple choice, yes/no, and Likert-scale items. An example question is, "Compared to one year ago, how would you rate your health in general now?" The SF-36 consists of eight scales (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health). Scores are converted into z-scores with a scale of 0-100 with 0 indicating the greatest level of disability and 100 the least.
Change from Baseline Parkinson's disease Quality of Life at 1-week post-intervention | 1-week post-intervention
  The Parkinson's Disease Quality of Life Questionnaire (PDQ-39) consists of 39 Likert-scale questions asking how often in the last month the participant experienced something due to having Parkinson's disease. An example question is, "Had difficulty doing leisure activities which you would like to do?" with response options for all questions being "never", "occasionally", "sometimes", "Often", and "always or cannot do at all". The overall score from the PDQ-39 can be used for a global assessment, and scores can also be broken down into the following individual scales: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communications and bodily discomfort.
Change from Baseline Healthy Lifestyle Behaviors at 1-week post-intervention | 1-week post-intervention
  The Lifestyle Profile II contains 52 Likert-scale items pertaining to healthy lifestyle behaviors in the areas of healthy eating, physical activity, spirituality, stress management, health responsibility, and interpersonal relations. Respondents are asked to indicate the frequency with which they engage in behaviors with the response options of "Never", "Sometimes", "Often", and "Routinely". An example question is, "Take some time for relaxation each day." Scores range from 52-208 and fall into the categories of poor (52-90), moderate (91-129), good (130-168), an excellent (169-208).
Change from Baseline Caregiver Burden at 1-week post-intervention | 1-week post-intervention
  The Zarit Burden Interview Short Form (ZBI-12) is designed to measure caregiver burden and consists of 12 Likert-scale items that ask respondents to if they feel a certain way "Never", "Rarely", "Sometimes", "Quite Frequently" or "Nearly Always". An example question is, "That because of the time you spend with your relative that you don't have enough time for yourself?" Scores range from 0-48 and are grouped into the categories of mild burden (0-10), mild to moderate burden (10-20), and high burden (>20).
Change from Baseline cognitive functioning at 1-week post-intervention | 1-week post-intervention
  The Montreal Cognitive Assessment (MoCA) is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Examples of questions include drawing a clock at ten past eleven and serial subtraction starting at 100. Scores on the MoCA range form 0-30 with a score of 26 or higher generally considered normal.
Change from Baseline Coping at 1-week post-intervention | 1-week post-intervention
  Ways of Coping is a 66 Likert-scale item instrument that assesses behaviors used to cope with everyday stressful encounters. Response options are "Not Used", "Used Somewhat", "Used Quite A Bit", and "Used A Great Deal". Respondents are asked to describe a stressful situation they experienced in the past week and to respond to each item asking to what extent they used that way of coping in that situation. Examples of items are, "Turned to work or substitute activity to take my mind off things" and "Found new faith". The items comprise eight scales: confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, and positive reappraisal.
Change from Baseline Depression Symptoms at 1-week post-intervention | 1-week post-intervention
  The Patient Health Questionnaire (PHQ-9) is used to measure depressive symptoms. The nine Likert-scale items have response options of, "Not at all", "Several days", "More than half the days", and "Nearly every day" and include questions such as, "Little interest or pleasure in doing things" and "Poor appetite or overeating." Scores range from 0-27 with 0 indicating no depression and five bands of scores ranges indicating minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe depression (20-27).
Change from Baseline Anxiety Symptoms at 1-week post-intervention | 1-week post-intervention
  The Generalized Anxiety Disorder (GAD-7) consists of seven Likert-scale items designed to measure anxiety. Response options are, "Not at all", "Several Days", "More than half the days", and "Nearly every day" and item examples are, "Trouble relaxing" and "Becoming easily annoyed or irritated". Scores range form 0-21 with scores of 8 or higher indicating a probable anxiety disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gonzalez, PhD, Principal Investigator — Stony Brook Medical Center
Locations (1):
- Stony Brook Medical Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No